CLINICAL TRIAL: NCT07407595
Title: Effect of Anticipated Pain on Corticospinal Excitability
Acronym: PACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universite du Littoral Cote d'Opale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A00353-46
Record Dates: First submitted 2025-12-17; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Nocebo Effect; Kinesiophobia
Keywords: Pain anticipation; Nocebo effect; Kinesiophobia; Corticospinal excitability; Transcranial magnetic stimulation
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups. Both groups receive the application of the same inert cream. The experimental group is informed that the cream is expected to induce pain, whereas the control group is informed that the cream is inactive.
Masking Description: A randomized number is allocated for all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Inert Cream (Neutral Information) (Other): Participants in this control arm receive the application of an inert cream on the forearm. They are informed that the cream is inactive and will not produce any sensation or effect. This arm serves as a control condition for the manipulation of pain anticipation, with identical procedures and measurements as the experimental arm, except for the information provided about the expected effects of the cream.
  Interventions: Other: Pain Expectation Manipulation
- Experimental Group - Inert Cream (Pain Expectation Information) (Experimental): Participants in this experimental arm receive the application of an inert cream on the forearm. They are informed that the cream is expected to induce painful sensations after a delay, with pain gradually increasing in intensity over time. This information is used to induce anticipation of pain without actual nociceptive stimulation. All procedures and measurements are identical to those of the control arm, except for the information provided about the expected effects of the cream.
  Interventions: Other: Pain Expectation Manipulation

INTERVENTIONS:
Other: Pain Expectation Manipulation — The intervention consists of an information-based manipulation designed to induce (or not induce) anticipation of pain. Participants receive the application of an inert cream on the forearm. Depending on group assignment, participants are informed either that the cream is inactive and will not produce any sensation, or that it is expected to produce painful sensations such as burning, stinging, or tingling, with onset approximately 10 minutes after application and a gradual increase in intensity over time, reaching a moderate to strong level of perceived pain. The cream itself has no active or sensory effects in any group. This intervention allows manipulation of pain expectation without inducing actual nociceptive stimulation.

SUMMARY:
The purpose of this study is to investigate how the anticipation of pain, in the absence of real pain, affects the excitability of the corticospinal pathway. Corticospinal excitability reflects how responsive the motor areas of the brain are when sending signals to muscles.

In this study, healthy adult participants will be randomly assigned to one of two groups. Both groups will receive the application of an inert cream on the forearm. Participants in the experimental group will be told that the cream may cause pain, while participants in the control group will be informed that the cream is completely inactive. In reality, the cream has no physical effect in either group. This design allows the researchers to isolate the effect of pain anticipation (a nocebo effect) without exposing participants to actual pain.

Corticospinal excitability will be measured using transcranial magnetic stimulation (TMS), a non-invasive technique that stimulates the motor cortex to assess brain-to-muscle communication. Measurements will be taken before and after the application of the cream.

In addition, psychological factors related to catastrophizing and fear of movement will be assessed using validated questionnaires, and physiological responses associated with stress will be measured through heart rate variability.

The main question this study aims to answer is whether anticipating pain, even without experiencing real pain, alters corticospinal excitability, and whether this effect is influenced by fear of movement and catastrophizing. By improving our understanding of how pain-related expectations affect brain function, this research may contribute to better strategies for preventing maladaptive motor changes associated with chronic pain.

DETAILED DESCRIPTION:
Pain-related processes involve not only sensory inputs but also cognitive and emotional factors such as expectation, fear, and anticipation. Anticipating pain can influence motor behavior and emotional responses even in the absence of actual nociceptive stimulation. These anticipatory mechanisms are thought to contribute to maladaptive motor adaptations and may play a role in the development and maintenance of chronic pain conditions. However, the neurophysiological effects of pain anticipation, independently of real pain, remain insufficiently understood.

The aim of this study is to examine the effect of pain anticipation on corticospinal excitability, a neurophysiological marker of motor cortex responsiveness and brain-to-muscle communication. Corticospinal excitability is assessed using transcranial magnetic stimulation (TMS) applied over the primary motor cortex. This non-invasive technique allows evaluation of motor pathway function through the elicitation of motor evoked potentials recorded from a target hand muscle.

To specifically investigate anticipation-related effects, the study uses an experimental paradigm designed to manipulate pain expectancy without inducing actual pain. In addition to neurophysiological measures, psychological factors related to fear of movement and physiological markers of autonomic nervous system activity are considered, as they may influence the impact of pain anticipation on motor system function.

Procedures :

After providing informed consent, participants take part in a single experimental session conducted in a laboratory setting. The session begins with baseline assessments designed to characterize neurophysiological, psychological, and autonomic parameters prior to any experimental manipulation.

Participants first complete self-report questionnaires assessing fear of movement, catastrophizing and pain-related avoidance beliefs (EKT-CF, PCS-CF and FACS-CF).

Baseline measurements of corticospinal excitability are then obtained using transcranial magnetic stimulation (TMS) applied over the primary motor cortex. The TMS will be used to establish the input-output (I/O) curves. Stimuli of variable intensity between the threshold value (or MT for motor threshold) and the maximum will be delivered. In total, about ten stimulation intensities will be tested, and for each stimulation intensity, ten stimuli will be delivered, allowing then to calculate the average of the MEPs in order to draw the I/O curves of each participant. The resulting motor evoked potentials to characterize global corticospinal responsiveness. As recalled by national and international recommendations, TMS is a noninvasive and painless technique whose use in the scientific literature is extremely abundant.

In parallel, baseline autonomic activity is recorded using heart rate variability measures.

Following baseline assessments, participants are randomly assigned to either an experimental group or a control group. In both groups, an inert cream is applied to a predefined area of the forearm. The manipulation differs only in the information provided to participants. Those assigned to the experimental group are informed that the cream is expected to induce painful sensations (such as burning or tingling) after an approximate delay of ten minutes, with the pain progressively increasing in intensity over time, whereas participants in the control group are informed that the cream is inactive and will not produce any sensation. In reality, the same inert cream is used for all participants. This procedure is designed to induce anticipation of pain in the experimental group without exposing participants to actual nociceptive stimulation.

Immediately after the application of the cream and the expectancy manipulation, corticospinal excitability is reassessed using the same TMS procedures as at baseline. Measurements are repeated to examine changes in motor system excitability associated with pain anticipation. Autonomic nervous system activity continues to be monitored throughout this phase.

To reinforce the anticipatory context, additional TMS measurements, using the same procedures, are performed around the time when participants in the experimental group are led to expect the onset of pain (approximatively 10 minutes after cream application). This allows assessment of corticospinal excitability during heightened anticipation, independently of any real sensory input.

At the end of the experimental session, participants are asked to report their perceived pain and level of apprehension during the study. A full debriefing is then conducted, during which the true purpose of the study and the use of expectancy manipulation are explained. Participants are given the opportunity to ask questions and withdraw their data if they wish.

The duration of the experimental session is estimated at 1h30min, distributed as follows: Information, eligibility and consent collection, questionnaires completion : 20 minutes; preparation of the experiment (installation of the electrodes, setting of the devices: 10 minutes; recordings: 1 hour).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* No current pain at the time of inclusion and no pain episode or injury associated with pain within the past 3 months.
* Ability to understand spoken and written French sufficient to follow study procedures.
* Written informed consent obtained prior to participation.
* Subjects affiliated with or receiving social security benefits

Exclusion Criteria:

* History of psychiatric disorders (including intellectual disability or severe cognitive, behavioral, or affective impairment) that could interfere with understanding the study or providing informed consent.
* History of neurological disorders, including epilepsy, stroke, brain or spinal cord surgery, or any neurological disease affecting motor or sensory function.

Inability to provide informed consent (e.g., dementia, significant hearing impairment, insufficient language proficiency).

* Any pain condition within the past 3 months, regardless of origin.
* Recent musculoskeletal injury or surgery within the past 3 months.
* Contraindications to transcranial magnetic stimulation (TMS), including a history of epilepsy or the presence of intracranial metallic objects, cochlear implants, or other non-removable metallic implants in or near the head.
* Use of analgesic or psychotropic medications.
* Individuals under legal guardianship or curatorship.
* Pregnant or breastfeeding women.
* Presence of a cardiac pacemaker or other implanted electronic medical device.
* Known allergy or history of skin reaction to any component of the inert cream used in the study (Medicafarm® Neutre Premium Longue Glisse).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in corticospinal excitability | During single session: baseline (pre-cream application), immediately post-cream application, and 10 minutes post-cream application
  Corticospinal excitability will be assessed using transcranial magnetic stimulation (TMS) applied over the primary motor cortex. Single magnetic pulses of increasing intensity will be delivered to construct input-output (I/O) recruitment curves for each participant at baseline, immediately after cream application, and 10 minutes after cream application. Stimulation intensity will be increased in 3-5% steps, and 10 stimuli will be delivered at each intensity level. Motor evoked potentials elicited by TMS will be recorded using surface electromyography from the first dorsal interosseous muscle of the hand.
  I/O curves will be modeled using a Boltzmann sigmoidal function, and the slope, plateau, and S50 parameters will be extracted. Changes in corticospinal excitability will be compared between groups across these time points.

SECONDARY OUTCOMES:
Fear-avoidance beliefs related to pain | Baseline
  Fear-avoidance beliefs will be assessed using the French-Canadian version Fear-Avoidance Components Scale (FACS-FR/CF), a self-report questionnaire designed to measure cognitive, emotional, and behavioral components of fear-avoidance related to pain. The scale includes items assessing pain-related fear, anxiety, catastrophic thinking, and avoidance behaviors.
  The FACS-FR/CF consists of 20 items rated on a Likert scale from 0 (strongly disagree) to 5 (strongly agree), yielding a total score ranging from 0 to 100. Higher scores indicate greater levels of fear-avoidance. Severity levels are commonly interpreted as subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80), and extreme (81-100).
Kinesiophobia | Baseline
  Kinesiophobia will be assessed using the French-Canadian version of the Tampa Kinesiophobia Questionnaire (EKT-CF). It takes the form of a self-reported questionnaire of 17 items using a Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree), with an acceptable degree of internal consistency (Cronbach's alpha = 0.71), satisfactory construct validity, and high sensitivity to change (intra-class correlation coefficient > 0.7). The total score is obtained by adding the value of the responses and is between 17 and 68. The value of 40/68 is considered as the threshold value at which kinesiophobia becomes significant.
Change in heart rate variability from Baseline | During the single study session, from the baseline resting period through completion of the TMS procedure (up to 60 minutes)
  Heart rate variability (HRV) will be assessed as an index of autonomic nervous system activity. R-R intervals will be continuously recorded throughout the single study session, starting with the baseline resting period and continuing through completion of the TMS procedure. Time-domain HRV parameters (e.g., mean heart rate, RMSSD) will be derived from the continuous recording to evaluate autonomic responses associated with pain anticipation.
Pain catastrophizing related to pain | Baseline
  Pain catastrophizing will be assessed using the French-Canadian version of the Pain Catastrophizing Scale (PCS-CF), a self-report questionnaire designed to measure catastrophic thoughts related to pain. The PCS-CF includes 13 items rated on a Likert scale from 0 ("not at all") to 4 ("all the time"), covering three dimensions: rumination, magnification, and helplessness. Item scores are summed to yield a total score ranging from 0 to 52, with higher scores indicating greater pain catastrophizing. A total score ≥30 has been proposed to identify clinically relevant levels of pain catastrophizing.
Change from baseline in intracortical inhibition and facilitation (SICI and SICF) | During single session: baseline (pre-cream application), immediately post-cream application, and 10 minutes post-cream application
  Intracortical inhibitory and facilitatory circuits will be assessed using paired-pulse transcranial magnetic stimulation applied over the primary motor cortex. A subthreshold conditioning stimulus (80% RMT) will be followed by a suprathreshold (120% RMT) test stimulus to quantify short-interval intracortical inhibition (SICI), whereas paired-pulse stimulation at facilitative interstimulus intervals will be used to quantify short-interval intracortical facilitation (SICF). These measures will be obtained for each participant at baseline, immediately after cream application, and 10 minutes after cream application. Motor evoked potentials elicited by TMS will be recorded using surface electromyography from the first dorsal interosseous muscle of the hand. SICI and SICF will be expressed as the ratio of conditioned to unconditioned MEP amplitude (e.g., % of test MEP).

OTHER OUTCOMES:
Brief Pain Inventory | Baseline
  Current pain status will be assessed using the Brief Pain Inventory, French version (BPI-FR), a self-report questionnaire widely used to evaluate pain severity and pain-related interference with daily activities. In this study, the BPI-FR is used to confirm the absence of clinically relevant pain at inclusion.
  The questionnaire includes 11 items: four items assessing pain intensity (worst, least, average, and current pain) and seven items assessing the extent to which pain interferes with daily functioning, mood, sleep, and social activities.
  Pain intensity and interference are rated on numeric scales ranging from 0 (no pain or no interference) to 10 (worst imaginable pain or complete interference). Higher scores indicate greater pain severity and impact.
Change from baseline in perceived apprehension | During the single study session: baseline (pre-cream application), immediately post-cream application, and 10 minutes post-cream application
  Perceived apprehension related to the experimental context will be assessed using a 0-10 numeric rating scale, where 0 indicates "no apprehension at all" and 10 indicates "the highest apprehension imaginable." Participants will rate their apprehension at predefined time points before and after the expectancy manipulation in order to evaluate changes in apprehension associated with the experimental instructions and procedures.
Change from baseline in perceived pain intensity | During the single study session: baseline (pre-cream application), immediately post-cream application, and 10 minutes post-cream application
  Perceived pain intensity will be assessed using a 0-10 numeric rating scale, where 0 indicates "no pain" and 10 indicates "the worst pain imaginable." Participants will rate perceived pain intensity at predefined time points before and after the expectancy manipulation in order to support the credibility of the experimental instructions and to explore whether pain anticipation may be associated with a perceived experience of pain in the absence of actual nociceptive stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurasport, Loos, Nord, France

IPD SHARING:
Plan to Share IPD: No